CLINICAL TRIAL: NCT00969722
Title: A Randomized Study of Monoclonal Antibody 3F8 Plus Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) Compared to 13-cis-Retinoic Acid Plus GM-CSF in High Risk Stage 4, Primary Refractory Neuroblastoma Patients
Brief Title: A Study of MAb-3F8 Plus Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) Versus 13-cis-Retinoic Acid (RA) Plus GM-CSF in Primary Refractory Neuroblastoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3F8-NB-201
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Primary Refractory Neuroblastoma
Keywords: Neuroblastoma; 3F8; Primary refractory
MeSH Terms: conditions — Neuroblastoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM I (Experimental): Intravenous MAb-3F8 plus Subcutaneous Granulocyte Macrophage Colony Stimulating Factor (GM-CSF)
  Interventions: Biological: MAb-3F8; Biological: Subcutaneous Granulocyte Macrophage Colony Stimulating Factor (GM-CSF)
- ARM II (Active Comparator): Oral 13-cis-Retinoic Acid (RA) plus Subcutaneous Granulocyte Macrophage Colony Stimulating Factor (GM-CSF)
  Interventions: Biological: Subcutaneous Granulocyte Macrophage Colony Stimulating Factor (GM-CSF); Biological: 13-cis-Retinoic Acid

INTERVENTIONS:
Biological: MAb-3F8
  Arms: ARM I
Biological: Subcutaneous Granulocyte Macrophage Colony Stimulating Factor (GM-CSF)
Biological: 13-cis-Retinoic Acid
  Arms: ARM II

SUMMARY:
This is a multicenter, randomized, controlled, open-label study. Patients meeting inclusion/exclusion criteria will be randomized (1:1) to receive two cycles of MAb-3F8 plus GM-CSF or RA plus GM-CSF. Patients who do not respond to their assigned treatment after two cycles may cross-over to receive the alternate treatment. Disease response and safety will be assessed in all patients after cycle 2 and after cycle 4.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of stage 4 neuroblastoma diagnosed in accordance with the International Neuroblastoma Staging System: either (a) histologic confirmation which may involve immunohistochemical, ultrastructural, and/or cytogenetic studies, or (b) elevated urinary catecholamines plus tumor cells/clumps in the bone marrow.
* Have evaluable disease or biopsy-proven stable disease in BM by histology or MIBG scan with MIBG-positive disease confined to the bone or bone marrow, plus urine catecholamine results, documented >3 weeks after conventional chemotherapy or >6 weeks after stem-cell transplantation. CT, MRI, or bone scan (if necessary) can be done at 2-3 weeks after conventional chemotherapy confirming that the chemotherapy, radiotherapy, and ABMT are not realistic curative options.
* Be between 18 months to 13 years old at diagnosis.
* Have recovered to grade 2 or better toxicities since their prior therapy.
* Must, if female of childbearing potential, be willing to use two forms of medically acceptable contraception (at least one barrier method) and have a negative pregnancy test at screening and monthly thereafter through the first four cycles of treatment.
* Have a performance score of at least 60 from Lansky Play Performance Scale if aged up to 16 years or at least 60 from Karnofsky Scale if aged more than 16 years.
* Have voluntarily agreed to participate.

Exclusion Criteria:

* Have measurable disease ≥ 1 cm assessed by CT or MRI.
* Have progressive disease (any new lesion; increase of any measurable lesion by >25%; or previous negative marrow positive for tumor).
* Have disease detectable in CNS (confirmed by CT or MRI of the brain at screening or within 8 weeks of randomization).
* Be receiving alternative therapy for the treatment of neuroblastoma, e.g. radiotherapy or chemotherapy within 3 weeks of randomization.
* Require additional therapy (such as radiotherapy) during the first two treatment cycles.
* Have detectable human anti-mouse antibody titers at screening.
* Have received prior anti-GD2 investigational therapies.
* Have a history of allergies to mouse proteins.
* Have an active infection requiring IV infusion of antibiotics.
* Be currently receiving long-term chronic treatment with immunosuppressive drugs such as cyclosporine, adrenocorticotropic hormone (ACTH), or systemic corticosteroids.

Ages: 18 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To compare the proportion of patients achieving a complete bone marrow response measured by an absence of histological evidence of bone marrow disease and by MIBG scan after two cycles of treatment. | two years

SECONDARY OUTCOMES:
A comparison in treatment arms for disease response as measured by CT/MRI scan and urine catecholamines, MIBG extent of disease scores, disease response in cross-over patients. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Peter E. Zage, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (15):
- United States (15):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Rady Children's Hospital of San Diego, San Diego, California
  - Georgetown Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital in Florida, St. Petersburg, Florida
  - LSU Health Sciences Center; Children's Hospital, New Orleans, Louisiana
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Childrens Hospital, Columbus, Ohio
  - University of Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - US Oncology, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - Vermont Cancer Center, Burlington, Vermont